CLINICAL TRIAL: NCT02471079
Title: TOxicity After Radiotherapy in breAst CancEr Survivors (ThORACeS) - A Retrospective Cohort Study
Acronym: THORACES
Status: Completed | Type: Observational
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Other Study IDs: RT2014-02
Record Dates: First submitted 2015-05-19; First posted 2015-06-15 (Estimated); Last update posted 2024-02-28 (Actual); Status verified 2024-02

CONDITIONS: Breast Cancer
Keywords: Radiation-induced health problems; Cardiovascular events; Lung toxicity
MeSH Terms: conditions — Breast Neoplasms | interventions — Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Radiation: Radiotherapy

SUMMARY:
Rationale:

The number of breast cancer (BC) patients at risk for long-term radiation-induced health problems is increasing, as their outcome is improving due to intensified treatment regimens, such as new systemic approaches and radiotherapy. Therefore, identifying BC survivors with the highest risk for radiation-induced health problems is crucial for developing strategies for primary and secondary prevention, which may contribute to healthy ageing.

ELIGIBILITY:
Inclusion Criteria:

* Female gender.
* Treated for stage I-III invasive adenocarcinoma of the breast or ductal carcinoma in situ (DCIS).
* Treated with curative breast-conserving surgery followed by radiotherapy of the breast, with or without irradiation of the regional lymph nodes.
* Start of radiotherapy is between 01-01-2005 and 31-12-2008.
* Available planning CT scan and dose distribution data of original breast cancer irradiation.

Exclusion Criteria:

* Any prior malignancy other than non-melanoma skin cancer or breast cancer.
* Prior radiotherapy treatments in the thoracic region.
* Treated with neoadjuvant chemotherapy.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult, female patients with stage I-III breast cancer, who were treated with breast-sparing surgery followed by radiation treatment.
Sampling Method: Non-Probability Sample
Enrollment: 706 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Number of participants with cardiovascular events in relation with the received heart radiation dose | At time of data collection: minimum at 7 years and maximum at 10 years after completion of radiation therapy
Number of participants with secondary malignancies in relation with the received radiation dose | At time of data collection: minimum at 7 years and maximum at 10 years after completion of radiation therapy
Number of participants with radiation pneumonitis in relation with the received lung radiation dose | At time of data collection: minimum at 7 years and maximum at 10 years after completion of radiation therapy
Number of participants with hypothyroidism in relation with the received radiation dose | At time of data collection: minimum at 7 years and maximum at 10 years after completion of radiation therapy

CONTACTS AND LOCATIONS:
Locations (1):
- University Medical Center Groningen, Groningen, Netherlands